CLINICAL TRIAL: NCT05040568
Title: A PHASE IB STUDY OF IMMUNOTHERAPY WITH EX VIVO PRE-ACTIVATED AND EXPANDED CB-NK CELLS IN COMBINATION WITH CETUXIMAB, IN COLORECTAL CANCER PATIENTS WITH MINIMAL RESIDUAL DISEASE (MRD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0076; NCI-2021-09411 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2021-08-24; First posted 2021-09-10 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Colon Cancer; Resected Stage
MeSH Terms: conditions — Colonic Neoplasms | interventions — Cetuximab; fludarabine phosphate; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cetuximab (Experimental): given to patients with high-risk colorectal cancer
  Interventions: Drug: Cetuximab; Drug: Expanded CB-NK cells; Drug: Fludarabine phosphate; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cetuximab — Given IV
  Other Names: C225; Erbituxâ"¢; IMC-C225; MOAB C225
Drug: Expanded CB-NK cells — Given IV
Drug: Fludarabine phosphate — Given IV
  Other Names: Fludarabine; FludaraÂ®
Drug: Cyclophosphamide — Given IV
  Other Names: CytoxanÂ®; NeosarÂ®

SUMMARY:
A study of immunotherapy with expanded CB-NK cells in combination with cetuximab, to evaluate activity against minimal residual disease in patients with colon cancer that have completed adjuvant treatment but are positive for ctDNA

DETAILED DESCRIPTION:
This is a Phase Ib clinical trial to evaluate the safety and activity of expanded CB-NK cells in combination with cetuximab in patients with high-risk CRC who have completed adjuvant chemotherapy but are still positive for MRD (see Figure 5). A total of 15 patients with stage II-III, and resected stage IV CRC and positivity for MRD will be enrolled. MRD is defined as the lack of radiographically evident disease, in the presence of ctDNA matching the original tumor mutations after adjuvant chemotherapy. The primary goal of the study is ctDNA clearance from the blood in these patients. After completing SOC surgery and adjuvant chemotherapy, patients will be tested for the persistence of blood ctDNA. Those who are ctDNA-positive will repeat a computed tomography (CT) scan and if the imaging shows no radiological evidence of disease, they will be eligible for the study screening.

Primary Objective:

• To evaluate the activity of the CB-NK infusion in combination with cetuximab in patients with resected colorectal cancer and positivity for minimal residual disease

Secondary Objective:

• To evaluate the efficacy of the CB-NK infusion in combination with cetuximab in patients with resected colorectal cancer and positivity for minimal residual disease

ELIGIBILITY:
Inclusion Criteria:

* Has high-risk stage II or stage III colorectal cancer and has completed standard-of-care treatment, including complete disease resection followed by standard-of-care adjuvant treatment and has no evidence of relapsing disease per the CT scan but has persistent ctDNA in the bloodstream; OR has resected stage IV colorectal cancer undergone with curative intent, has completed standard-of-care adjuvant- and/or neo-adjuvant treatment, and has no evidence of residual disease per the CT scan but has persistent ctDNA in the bloodstream.
* Has signed the Informed Consent Form
* Is age ≥ 18 years
* Is able to comply with the study protocol, in the investigator's judgment
* Has ECOG performance status of 0-1
* Has adequate hematologic and end-organ function defined by the following laboratory test results obtained within 28 days prior to initiation of study treatment:

  * Absolute neutrophil count (ANC) ≥ 1,500/mm3 without granulocyte colony-stimulating factor support
  * Lymphocyte count ≥ 500/mm3
  * Platelet count ≥ 100,000/mm3 without transfusion
  * White blood cell count ≥ 2,500/mm3
  * Hemoglobin ≥ 9.0 g/dL o Patients may be transfused to meet this criterion.
  * Aspartate transaminase (AST), alanine transaminase (ALT), and alkaline phosphatase ≥ 2.5 x upper limit of normal (ULN), with the following exceptions:

    * For patients with documented liver metastases: AST and ALT ≤ 5 x ULN
    * For patients with documented liver or bone metastases: alkaline phosphatase ≤ 5 x ULN
  * Serum bilirubin ≤ 1.5 x ULN with the following exception:

    o For patients with known Gilbert disease: serum bilirubin level ≤ 3 x ULN
  * Serum creatinine ≤ 1.5 x ULN
  * Serum albumin ≥ 2.5 g/dL
  * For patients not receiving therapeutic anticoagulation: international normalized ratio (INR) or activated partial thromboplastin time (aPTT) ≤1.5 x ULN
  * Adequate cardiac function

    * Baseline EKG and echocardiogram (ECHO) within normal limits
* For women and men for childbearing potential: agreement to use a contraceptive method with a failure rate of <1% per year or remain abstinent (refrain from heterosexual intercourse) during the treatment period and for 6 months after the last dose of study treatment

  * A woman is considered to be of childbearing potential if she is premenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
  * Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, barrier method, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

* Received treatment for the studied cancer within 28 days prior to initiation of study treatment
* Received treatment with an investigational therapy within 28 days prior to initiation of study treatment
* Has a history of severe allergic-, anaphylactic-, or other hypersensitivity reactions to chimeric- or humanized antibodies or fusion proteins
* Has a known hypersensitivity to biopharmaceutical agents produced in Chinese hamster ovary cells
* Has a known allergy or hypersensitivity to any component of the expanded CB-NK cells formulation
* Has a known allergy or hypersensitivity to any component of the cetuximab formulation
* Has active- or a history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

  • Patients with a history of autoimmune-related hypothyroidism who are on thyroid- replacement hormone are eligible for the study.
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    * Rash must cover <10% of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
    * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months
* Had prior allogeneic stem cell or solid organ transplantation
* Has history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan

  • History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Had a positive HIV test at screening
* Has active hepatitis B virus (HBV) infection (chronic or acute), defined as having a positive hepatitis B surface antigen (HBsAg) test at screening

  • Patients with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive total hepatitis B core antibody (HBcAb) test and negative HBV DNA test at screening, are eligible for the study.
* Has active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test followed by a positive HCV RNA test at screening

  • The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
* Has active tuberculosis
* Had a severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Had treatment with therapeutic oral or intravenous (IV) antibiotics within 2 weeks prior to initiation of study treatment

  • Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Has significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction, unstable arrhythmia, unstable angina, or cerebrovascular accident within 3 months prior to initiation of study treatment
* Had a major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipates needing a major surgical procedure during the course of the study
* Received treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipates needing such a vaccine during the course of the study, or up to 5 months following the anticipated dose of expanded CB-NK cells.
* Had a malignancy other than the disease under study within 5 years prior to receipt of expanded CB-NK cell therapy.

  • Allowed are (1) those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ treated surgically with curative intent); or (2) those undergoing active surveillance per standard-of-care management (e.g., chronic lymphocytic leukemia Rai Stage 0)
* Has any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Had treatment with any immune checkpoint blockade therapy, including antiCTLA-4, antiPD-1, or antiPD-L1 therapeutic antibodies, within 4 weeks or five half-lives of the drug prior to initiation of this study
* Received treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2) within 4 weeks or five half-lives of the drug (whichever is longer) prior to initiation of study treatment
* Received treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and antiTNF- agents) within 2 weeks prior to initiation of study treatment, or anticipates needing systemic immunosuppressive medication during the course of the study, with the following exceptions:

  * Patients who received low-dose immunosuppressant medication are eligible for the study.
  * Patients with active immunological disease requiring more than 10 mg of steroids daily are eligible for the study.
  * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* Is pregnant or breastfeeding, or intends to become pregnant during the study • Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
The activity of the CB-NK infusion in combination with cetuximab in patients with resected colorectal cancer and positivity for minimal residual disease | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Maria Morelli, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-10-23): https://cdn.clinicaltrials.gov/large-docs/68/NCT05040568/ICF_001.pdf